CLINICAL TRIAL: NCT02378324
Title: Effect of Fee on Attendance in Cervical Cancer Screening-results From ScreenFee a Swedish Population Based Randomised Trial
Brief Title: Effect of Fee on Attendance in Cervical Cancer Screening
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Göteborg University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Screening
Other Study IDs: ScreenFee
Record Dates: First submitted 2015-01-05; First posted 2015-03-04 (Estimated); Last update posted 2015-03-04 (Estimated); Status verified 2015-02

CONDITIONS: Cervical Dysplasia
Keywords: Attendance; Screening without fee
MeSH Terms: conditions — Uterine Cervical Dysplasia | interventions — Mass Screening; Fees and Charges

STUDY DESIGN:
Who Masked: Care Provider
Oversight: Data Monitoring Committee: No

ARMS (2):
- Intervention and control (Active Comparator): Intervention arm: screening without fee.
  Interventions: Other: Screening without fee
- Control group (No Intervention): Control arm: screening with the regular fee, 100SEK.

INTERVENTIONS:
Other: Screening without fee — All women in three districts in Gothenburg, Sweden, that were eligible for invitation in the regular screening program were individually randomized by computer program in two parallel arms 1:1.
  Arms: Intervention and control

SUMMARY:
Several reasons can explain non-attendance in cervical cancer screening. In low resource settings the attendance is even lower. The effect of fee as contributing reason of non attendance has not been studied before why the investigators decided to study this in a low resource setting as a randomised trial.

DETAILED DESCRIPTION:
Non-attendance in the cervical cancer screening programme is the most important factors why Swedish women contract the disease. Low attendance rate is observed in districts with low socioeconomic resources. Several reasons can explain this, including the existence of a fee. A low attendance rate in low resource districts is also noticed in Gothenburg, Sweden. After multiple interventions the coverage has slightly increased. None of the interventions included the aspect of the fee. The investigators decided to study the effect of fee abolishment in a randomized control trial emanating from the regular cervical cancer-screening program. Method: Randomized Control Trial (RCT). Women in low resource areas of Gothenburg, due for screening, January-July 2013, were randomised to receive an offer of a free test or receiving the regular invitation stating the regular fee of 100 Swedish kronor (SEK) (≈11 €). Power calculation has shown 80 % power to detect an increase in participation of 20% at 1972 participants.

ELIGIBILITY:
Inclusion Criteria:

* All women in the designated geographical area, consecutively enrolled in planned screening according to standard routine. I.e women are invited if they are between 23 and 60 years of age and don't have a pap smear registered the last three or five years according to age.

Exclusion Criteria:

* None

Ages: 23 Years to 60 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 3124 (Actual)
Dates: Start 2013-01; Primary Completion 2013-07 (Actual); Study Completion 2013-07 (Actual)

PRIMARY OUTCOMES:
Difference in attendance | 6 months
  Information from the database regarding study arm was linked, via citizen unique personal number, to the National Cervical Screening Quality Register. From this database aggregated information of attendance was extracted. The effect of the intervention on attendance was calculated as relative risks.

SECONDARY OUTCOMES:
Differences in attendance stratified for age groups, home districts and previous pap smear history. | 6 months
  Before analysing the results of which kind of invitation the woman got, age group, previous pap smear history and district, all personal information was anonymized.

CONTACTS AND LOCATIONS:
Overall Officials: Björn Strander, PhD, Study Director — Regional Cancer Center West

REFERENCES:
- [Background] Broberg G, Jonasson JM, Ellis J, Gyrd-Hansen D, Anjemark B, Glantz A, Soderberg L, Ryd ML, Holtenman M, Milsom I, Strander B. Increasing participation in cervical cancer screening: telephone contact with long-term non-attendees in Sweden. Results from RACOMIP, a randomized controlled trial. Int J Cancer. 2013 Jul;133(1):164-71. doi: 10.1002/ijc.27985. Epub 2013 Jan 10. PMID 23233356
- [Background] Andrae B, Kemetli L, Sparen P, Silfverdal L, Strander B, Ryd W, Dillner J, Tornberg S. Screening-preventable cervical cancer risks: evidence from a nationwide audit in Sweden. J Natl Cancer Inst. 2008 May 7;100(9):622-9. doi: 10.1093/jnci/djn099. Epub 2008 Apr 29. PMID 18445828
- [Background] Segnan N, Senore C, Giordano L, Ponti A, Ronco G. Promoting participation in a population screening program for breast and cervical cancer: a randomized trial of different invitation strategies. Tumori. 1998 May-Jun;84(3):348-53. doi: 10.1177/030089169808400307. PMID 9678615
- [Background] Eaker S, Adami HO, Granath F, Wilander E, Sparen P. A large population-based randomized controlled trial to increase attendance at screening for cervical cancer. Cancer Epidemiol Biomarkers Prev. 2004 Mar;13(3):346-54. PMID 15006907
- [Background] Broberg G, Gyrd-Hansen D, Miao Jonasson J, Ryd ML, Holtenman M, Milsom I, Strander B. Increasing participation in cervical cancer screening: offering a HPV self-test to long-term non-attendees as part of RACOMIP, a Swedish randomized controlled trial. Int J Cancer. 2014 May 1;134(9):2223-30. doi: 10.1002/ijc.28545. Epub 2013 Oct 31. PMID 24127304
- [Background] Wikstrom I, Lindell M, Sanner K, Wilander E. Self-sampling and HPV testing or ordinary Pap-smear in women not regularly attending screening: a randomised study. Br J Cancer. 2011 Jul 26;105(3):337-9. doi: 10.1038/bjc.2011.236. Epub 2011 Jul 5. PMID 21730977
- [Background] Idestrom M, Milsom I, Andersson-Ellstrom A. Knowledge and attitudes about the Pap-smear screening program: a population-based study of women aged 20-59 years. Acta Obstet Gynecol Scand. 2002 Oct;81(10):962-7. doi: 10.1080/j.1600-0412.2002.811011.x. PMID 12366488
- [Derived] Alfonzo E, Andersson Ellstrom A, Nemes S, Strander B. Effect of Fee on Cervical Cancer Screening Attendance--ScreenFee, a Swedish Population-Based Randomised Trial. PLoS One. 2016 Mar 17;11(3):e0150888. doi: 10.1371/journal.pone.0150888. eCollection 2016. PMID 26986848